CLINICAL TRIAL: NCT06820905
Title: Hyperinflammation and Hyperferritinemia in Critically Ill Patients: a Retrospective Observational Single-center Analysis
Brief Title: Hyperinflammation and Hyperferritinemia in Critically Ill Patients
Acronym: HYFER
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Thomas Karvunidis, Principal investigator, Charles University, Czech Republic
Other Study IDs: HYFER_2025
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Sepsis; Hyperferritinemia; Hyperinflammatory Syndrome
Keywords: criticall illness; sepsis; ferritin; hyperinflammatory syndrome; sepsis phenotype
MeSH Terms: conditions — Critical Illness; Sepsis; Hyperferritinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- critically ill patients: critically ill patients admitted to ICU between 01.01.2020 and 31.12.2024

SUMMARY:
Analysing trajectory of critically ill patients with signs of hyperinflammation

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* admission between 01.01.2020 and 31.12.2024 (5yrs)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients; mix-cases medical ICU population
Sampling Method: Non-Probability Sample
Enrollment: 1962 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
hyperferritinemia | 2025
  trajectory of critically ill patients with significant hyperferritinemia and with regard to its dynamics; ferritin value cutt-off

SECONDARY OUTCOMES:
etiology and association of hyperferritinemia | 2025
  etiology and association of hyperferritinemia with infectioius a non-infectious diseases/conditions
mortality a morbidity | 2025
  mortality a morbidity of patients with significant hyperferritinemia
treatment strategy | 2025
  association of hyperferritinemia and treatment strategy
stratification | 2025
  patient stratification according to hyperferritinemia/hyperinflammation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Karvunidis, MD, PhD, Principal Investigator — Faculty of Medicine and Teaching Hospital, Charles University, Pilsen, Czech Republic
Locations (1):
- Faculty of Medicine and Teaching Hospital, Charles University, Pilsen, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR